CLINICAL TRIAL: NCT06074211
Title: Development and Incorporation of Safe Sleep Education Into m-Health Technology for the Pediatric Emergency Department
Brief Title: Incorporation of Safe Sleep Education Into m-Health Technology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American SIDS Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00362756
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Sudden Infant Death
MeSH Terms: conditions — Sudden Infant Death | interventions — Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe Sleep Education (Experimental): The intervention group will receive safe sleep education via the Safety in Seconds mobile app.
  Interventions: Behavioral: Safety in Seconds mobile app: Safe Sleep Education
- Car seat safety (Active Comparator): The attention matched control group will receive car seat safety education via the Safety in Seconds mobile app.
  Interventions: Behavioral: Safety in Seconds mobile app: Car Seat Safety Education

INTERVENTIONS:
Behavioral: Safety in Seconds mobile app: Safe Sleep Education — The Safety in Seconds mobile app is a platform previously developed to deliver targeted injury prevention education. This intervention will be testing the effectiveness of a newly developed educational module on safe sleep education.
  Arms: Safe Sleep Education
Behavioral: Safety in Seconds mobile app: Car Seat Safety Education — The Safety in Seconds mobile app is a platform previously developed to deliver targeted injury prevention education, including fire and car seat safety.
  Arms: Car seat safety

SUMMARY:
Sudden Unexplained Infant Death (SUID) is the leading cause of death in infants age 28 days to 1 year. Protective factors, such as supine positioning, firm sleep surface, breastfeeding, pacifier use, elimination of soft objects from the sleep space, and avoidance of tobacco, alcohol, and illicit drugs have been shown to decrease the risk. The American Academy of Pediatrics recommends that healthcare providers model and convey safe sleep practices during patient encounters. Pediatric emergency departments (PED) serve as front-line contact for populations at greatest risk for SUID, however few interventions have been tested in the PED setting. M- Health (mobile health) apps have previously demonstrated the ability to deliver safety education to parents and are well suited for use in the PED given limited clinician time and long wait times. Safety in Seconds (SIS) is a theory based, m-Health injury prevention tool focused on care seat safety and fire safety with previously demonstrated effectiveness in an NIH-funded randomized trial. This study aims to add safe sleep education into the SIS, and subsequently disseminate the app in the PED setting. Integration of safe sleep education into SIS represents an opportunity to increase safe sleep knowledge and practices through a proven effective m-Health intervention. This study addresses this potential by incorporating a previously developed, theory-driven and evidence-based safe sleep education into the SIS app and testing the feasibility of deployment in the PED.

DETAILED DESCRIPTION:
More than 3500 children die annually in the US from Sudden Unexplained Infant Death (SUID) and sleep-related causes. Among the groups at highest risk for unsafe sleep behaviors and sleep-related infant mortality are racial and ethnic minorities, young mothers, and parents with substance use disorders. Safe sleep education is of great importance for the local community as infant mortality rates are notably high in Baltimore City. In 2017, Baltimore City's infant mortality rate was 1.3 times that of the state of Maryland and 1.5 times greater than the U.S. average. Of these deaths, 16.3% were related to sleep in Baltimore City compared to only 6.5% in the U.S. as a whole. Although attempts at integrating safe sleep education into health care visits have been met with varying success, the investigators have developed a theory- driven and evidence-based safe sleep intervention that increased safe sleep knowledge and practices.

Given that rates of sleep-related deaths have plateaued in the past decade, new prevention strategies are needed. For instance, strategic use of technology-based approaches as well as targeted efforts in the pediatric emergency department (PED) setting merit consideration for several reasons. First, smartphones and mobile applications provide additional opportunities to disseminate health education to parents. M-Health (mobile health) education apps have demonstrated the ability to deliver safety education. However, the efficacy of mobile applications for increasing adherence to safe sleep recommendations has not been tested. Second, there is a growing emphasis on the need for prevention and health education in the emergency department. The emergency department is also particularly well suited for the employment of technology-based interventions, as clinicians have limited time to provide education while patients often face long wait times. In the Johns Hopkins PED, previous research has demonstrated high smartphone use, and acceptability of such interventions. Further, many SUID cases had in emergency departments visits prior to death, which represents a missed opportunity to intervene and educate families about safe sleep, making safe sleep education in the PED imperative. Finally, many urban PEDs, serve a population at high risk for infant mortality due to sociodemographic factors.

To address these gaps and needs, this study proposes to adapt the Safety in Seconds (SIS) app to include safe sleep content and pilot test in the PED setting. The SIS app is a theory-based, m-Health tool that has been previously tested in the PED in an NIH-funded randomized trial that demonstrated its efficacy in improving appropriate car seat and smoke alarm knowledge and use. This app provides computer-generated, tailored messages to parents. There are three steps involved in the tool: (1) assessment; (2) data processing; and (3) feedback. Parents complete an assessment in the app and the answers are processed by a computer program to link each answer to specific theory-driven messages that are responsive to parents' reported beliefs and practices. These messages are used to produce a computer-generated, tailored report with persuasive and informative messages about safety topics. Building on this SIS app with proven effectiveness, the goal of this project is to incorporate evidence based, previously developed safe sleep education into the app and encourage implementation of safe sleep practices among families presenting to the PED.

Aim 1: Digitize existing educational content on infant safe sleep recommendations and incorporate into the SIS app (following the previously utilized process for the current app content on car seat safety and fire safety).

Aim 2: Pilot test the updated m-Health tool - SIS 2.0 - which incorporates new infant safe sleep content (from Aim 1) with existing injury prevention content on child passenger safety and fire safety. Feedback will be obtained from parents through follow-up surveys and interviews. Hypothesis: use of the SIS app for provision of safe sleep education will be effective in conveying this education.

ELIGIBILITY:
Inclusion Criteria:

* English speaking caregivers over 18 of infants age 0-4 months
* Use a smart phone

Exclusion Criteria:

* Non English speaking
* Under 18 years of age or unable to consent for themselves
* High acuity, critical care needs of infant patient that would limit participation during initial PED visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Safe sleep behaviors as assessed by survey developed by study team | Baseline, 1 month
  Safe sleep behaviors will be measured by the number of participants who adapt safe sleep behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Howard, MD, MSc, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Moon RY, Carlin RF, Hand I; TASK FORCE ON SUDDEN INFANT DEATH SYNDROME AND THE COMMITTEE ON FETUS AND NEWBORN. Sleep-Related Infant Deaths: Updated 2022 Recommendations for Reducing Infant Deaths in the Sleep Environment. Pediatrics. 2022 Jul 1;150(1):e2022057990. doi: 10.1542/peds.2022-057990. PMID 35726558
- [Background] Allen K, Anderson TM, Chajewska U, Ramirez JM, Mitchell EA. Factors associated with age of death in sudden unexpected infant death. Acta Paediatr. 2021 Jan;110(1):174-183. doi: 10.1111/apa.15308. Epub 2020 May 12. PMID 32304589
- [Background] Carlin RF, Moon RY. Risk Factors, Protective Factors, and Current Recommendations to Reduce Sudden Infant Death Syndrome: A Review. JAMA Pediatr. 2017 Feb 1;171(2):175-180. doi: 10.1001/jamapediatrics.2016.3345. PMID 27918760
- [Background] Canter J, Rao V, Patrick PA, Alpan G, Altman RL. The impact of a hospital-based educational video on maternal perceptions and planned practices of infant safe sleep. J Spec Pediatr Nurs. 2015 Jul;20(3):187-92. doi: 10.1111/jspn.12114. Epub 2015 Apr 21. PMID 25898856
- [Background] McDonald EM, Davani A, Price A, Mahoney P, Shields W, Musci RJ, Solomon BS, Stuart EA, Gielen AC. Health education intervention promoting infant safe sleep in paediatric primary care: randomised controlled trial. Inj Prev. 2019 Jun;25(3):146-151. doi: 10.1136/injuryprev-2017-042421. Epub 2017 Sep 22. PMID 28939661
- [Background] Gielen AC, McKenzie LB, McDonald EM, Shields WC, Wang MC, Cheng YJ, Weaver NL, Walker AR. Using a computer kiosk to promote child safety: results of a randomized, controlled trial in an urban pediatric emergency department. Pediatrics. 2007 Aug;120(2):330-9. doi: 10.1542/peds.2006-2703. PMID 17671059
- [Background] Nansel TR, Weaver N, Donlin M, Jacobsen H, Kreuter MW, Simons-Morton B. Baby, Be Safe: the effect of tailored communications for pediatric injury prevention provided in a primary care setting. Patient Educ Couns. 2002 Mar;46(3):175-90. doi: 10.1016/s0738-3991(01)00211-7. PMID 11932115